CLINICAL TRIAL: NCT05064475
Title: Correlation Between Petct Based Quantitative Parameters and CA 15.3 in Suspected Recurrent Breast Cancer
Brief Title: Correlation Between PET/CT Parameters and Tumor Markers in Recurrent Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SASamy, Salma Ahmed Samy anwar, Assiut University
Other Study IDs: Cpetptmrbc
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recurrent breast cancer patients with elevated tumor markers: PET/CT is the functional imaging tool that can measure increased glucose metabolism in cancer cells by using 18F-FDG. Its ability to identify tumor recurrence before detection of morphologic changes in conventional imaging reflecting its importance in detecting BC recurrence in asymptomatic patients with high tumor markers and negative results of radiological imaging. 18F-FDG PET/CT is frequently used for BC evaluation. However, data on its value in evaluating BC recurrence in patients with elevated tumor markers are limited and unclear
  Interventions: Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/CT — Patients with previous breast cancer, already treated and with clinical or biochemical suspicion of disease relapse. All patients will underwent 18F-fluorodeoxyglucose (FDG) PET/CT. In all patients, the value of CA 15.3 was compared to PET/CT. The final diagnosis of relapse will be derived from histopathological sampling As much as possible or radiological follow up for at least 6 months will be compared with PET/CT results.

SUMMARY:
Worldwide, breast cancer (BC) is the most frequent type of cancer in women yet, it is associated with relatively lower mortality rates, as it ranks fifth in cancer-related deaths overall, which is attributed to evolution in the treatment of recurrent and metastatic lesions, especially when these lesions were detected early . BC recurrence can occur even 15 years after primary treatment.

DETAILED DESCRIPTION:
life-long routine monitoring is mandatory. Although histopathologic confirmation is the definitive diagnostic method for BC recurrence, it is not always easy to perform as in cases with deeply located or very small-size lesions, or lesion too close to organs or great vessels, making sampling either inaccessible or hazardous. BC recurrence can be assessed using morphological imaging studies or tumor markers. Mammography, ultrasound (US), computed tomography (CT), and magnetic resonance imaging (MRI) are currently the most commonly used morphological imaging methods for detecting breast cancer recurrence. However, both of the two modalities have some restrictions.

Cancer antigen 15-3 (CA 15-3) and carcinoembryonic antigen (CEA) are two tumor markers that are frequently used in the monitoring of BC patients . However, the findings of many studies on these markers in BC follow-up are conflicting.

The introduction of integrated 2-deoxy-2-[18 F] fluoro-D-glucose (18FDG) positron emission tomography (PET) computed tomography (CT), known as PET/CT, has become a helpful tool for this purpose.

PET/CT is the functional imaging tool that can measure increased glucose metabolism in cancer cells by using 18F-FDG. Its ability to identify tumor recurrence before detection of morphologic changes in conventional imaging reflecting its importance in detecting BC recurrence in asymptomatic patients with high tumor markers and negative results of radiological imaging. 18F-FDG PET/CT is frequently used for BC evaluation. However, data on its value in evaluating BC recurrence in patients with elevated tumor markers are limited and unclear

ELIGIBILITY:
Inclusion Criteria:

* female patient with pathologically proved breast cancer who will be referred to do PET\CT imaging at the nuclear medicine unit, Assiut university hospital due to suspicion of recurrence based on elevated level of tumor marker in the period between October 2021 until the end of the study .

Exclusion Criteria:

* patients with newly diagnosed BC patients with early stages of BC BC patients with normal serum level of tumor markers

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: female patient with pathologically proved breast cancer who will be referred to do PET\CT imaging at the nuclear medicine unit, Assiut university hospital due to suspicion of recurrence based on elevated level of tumor marker
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
identification of recurrence | 2 years
  correlation between PET/CT parameters and the serum level of tumour markers in suspected recurrent BC as well as finding the best cut-off value of tumor markers that can be used in the identification of recurrence

REFERENCES:
- [Background] Ayala de la Pena F, Ortiz-Munoz B, Quintanar-Verduguez T, Santotoribio JD, de la Cruz S, Trape-Pujol J, Galve-Calvo E, Auge-Fradera JM, Garcia-Gomez J, Gonzalez-Hernandez A. Consensus of the Spanish society of laboratory medicine and the Spanish society of medical oncology on the methodology and criteria for evaluation of circulating tumour markers in breast cancer. Clin Transl Oncol. 2021 Jul;23(7):1272-1280. doi: 10.1007/s12094-020-02529-x. Epub 2021 Feb 7. PMID 33550504
- [Background] Liu C, Chen M, Shi Y. Downregulation of hsa_circ_0006220 and its correlation with clinicopathological factors in human breast cancer. Gland Surg. 2021 Feb;10(2):816-825. doi: 10.21037/gs-21-42. PMID 33708563
- [Background] Khushk M, Khan A, Rehman A, Sheraz S, Tunio YM, Rehman K, Rehman D, Ahmed M, Abbas K, Khan ME. The Role of Tumor Markers: Carcinoembryonic Antigen and Cancer Antigen 15-3 in Patients With Breast Cancer. Cureus. 2021 Jul 10;13(7):e16298. doi: 10.7759/cureus.16298. eCollection 2021 Jul. PMID 34405063
- [Background] Stergiou N, Nagel J, Pektor S, Heimes AS, Jakel J, Brenner W, Schmidt M, Miederer M, Kunz H, Roesch F, Schmitt E. Evaluation of a novel monoclonal antibody against tumor-associated MUC1 for diagnosis and prognosis of breast cancer. Int J Med Sci. 2019 Aug 14;16(9):1188-1198. doi: 10.7150/ijms.35452. eCollection 2019. PMID 31588183